CLINICAL TRIAL: NCT00845208
Title: Network and Contingency Management for Alcohol Treatment
Brief Title: Network Support for Treatment of Alcohol Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Mark Litt, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AA12827; R01AA012827 (NIH); 1R01AA012827 (NIH)
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Alcohol Dependence
Keywords: Network Support; AA; Contingency Management
MeSH Terms: conditions — Alcoholism | interventions — Support Vector Machine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Case Management (Active Comparator)
  Interventions: Behavioral: Network Support
- Network Support (Experimental): 12 Weekly sessions intended to help patients change their social networks to be more supportive of abstinence
  Interventions: Behavioral: Network Support
- Network Support + Contingency Mgmnt (Experimental): 12 weekly sessions intended to help patients change their social networks to be more supportive of abstinence. Contingency management component added to reinforce efforts to make network changes.
  Interventions: Behavioral: Network Support

INTERVENTIONS:
Behavioral: Network Support — 12 Weekly sessions intended to help patients change their social networks to be more supportive of abstinence

SUMMARY:
Relapse is the most serious problem in alcoholism treatment. The overall aim of the present study was to determine if a treatment directed at changing the patient's social network, from one that reinforces drinking behavior to one that reinforces sobriety, can create the conditions necessary for long-term treatment success. In addition, we intended to determine if explicit reinforcement for this change of social network (Contingency Management or ContM) would be more effective than the same network support intervention without contingent reinforcement for change.

ELIGIBILITY:
Inclusion Criteria:

* meet DSM-IV criteria for Alcohol Dependence
* at least 18 years old
* Willing to accept random assignment to treatment conditions

Exclusion Criteria:

* acute medical or psychiatric problems that require inpatient treatment
* reading ability below the fifth grade level
* lack of reliable transportation to the treatment site
* excessive commuting distance to site
* current dependence on drugs (except marijuana)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2002-03; Primary Completion 2007-10 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Proportion Days Abstinent | Every 3 months out to 2 years

SECONDARY OUTCOMES:
Network Support for Abstinence | every 6 months out to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Litt, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut health Center, Farmington, Connecticut, United States

REFERENCES:
- [Result] Litt MD, Kadden RM, Kabela-Cormier E, Petry N. Changing network support for drinking: initial findings from the network support project. J Consult Clin Psychol. 2007 Aug;75(4):542-55. doi: 10.1037/0022-006X.75.4.542. PMID 17663609
- [Result] Litt MD, Kadden RM, Kabela-Cormier E, Petry NM. Changing network support for drinking: network support project 2-year follow-up. J Consult Clin Psychol. 2009 Apr;77(2):229-42. doi: 10.1037/a0015252. PMID 19309183
- [Derived] Litt MD, Kadden RM, Tennen H. Treatment response and non-response in CBT and Network Support for alcohol disorders: targeted mechanisms and common factors. Addiction. 2018 Aug;113(8):1407-1417. doi: 10.1111/add.14224. Epub 2018 Apr 20. PMID 29575339